CLINICAL TRIAL: NCT04825925
Title: Drug-eluting Beads Bronchial Arterial Chemoembolization in Stage II-III Non-small-cell Lung Cancer Patients Failed, Refused or Ineligible to Receive Standard Treatments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20210168A
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DEB-BACE (Experimental)
  Interventions: Device: DEB-BACE(Drug-eluting beads bronchial arterial chemoembolization)

INTERVENTIONS:
Device: DEB-BACE(Drug-eluting beads bronchial arterial chemoembolization) — Bronchial arteriography was performed to find tumor-feeding artery. After the catheter had been inserted into the tumor-feeding artery, the Platinum was infused. BAI (Bronchial Arterial Infusion ) chemotherapy was followed by DEB-BACE(Drug-eluting beads bronchial arterial chemoembolization); the CalliSpheres loaded with Vinorelbine were infused into the tumor-feeding arteries until stasis or near-stasis of blood flow in the vessel was observed.

SUMMARY:
This is a multicenter, prospective, single-arm clinical study to determine the efficacy and safety of Drug-eluting beads bronchial arterial chemoembolization（DEB-BACE） in stage II-III NSCLC patients who failed, refused or ineligible to receive standard treatments

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years old, of any sex;
2. Patients who have histopathological proof of NSCLC according to the standard of diagnosis and treatment of primary lung cancer（V2018）;
3. Confirmed TNM stage is II-III of NSCLC;
4. Patients who were failed, refused or assessed ineligible by MDT to receive conventional Second-Line treatments (surgery, chemoradiotherapy, targeted and immunotherapy)；
5. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0-2;
6. Life expectancy of > 3 months;
7. Patients volunteered to participate in this study and signed informed consent, with good compliance;

Exclusion Criteria:

1. Patients received interventional therapy (I seeds implantation, Ablation, BACE) before;
2. A history combined with other malignant tumors and not cured;
3. WBC<3×109/L、LYM<1.5×109/L、NLR≥3、PLT<50×109/L、HGB<90 g/L;
4. Insufficient of liver and renal function (Cr>176.8 µmol/L; AST and/or ALT>2 folds of normal value)；
5. Combined with uncorrectable coagulation dysfunction or active massive hemoptysis;
6. Combined with active affection and need antibiotic treatment;
7. Uncontrollable hypertension, diabetes, cardiovascular disease with obvious symptoms;
8. Known to be hypersensitive to contrast agent;
9. Pregnant or breastfeeding women;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Time from the first DEB-BACE treatment to either radiological progression after the second DEB-BACE treatment or death, up to 36 months
  Time from the first DEB-BACE treatment to either radiological progression after the second DEB-BACE treatment or death

SECONDARY OUTCOMES:
Objective response rate (ORR) | 1, 3, 6 months after the first DEB-BACE treatment, up to death or 36months
  Proportion of patients with reduction in stable in tumor burden of a predefined amount
Disease control rate (DCR) | 1, 3, 6 months after the first DEB-BACE treatment, up to death or 36months
  Proportion of patients with reduction or keeping in stable in tumor burden of a predefined amount
Overall survival (OS) | Time from the first DEB-BACE treatment to death or up to 36 months
  Time from the first DEB-BACE treatment to death from any cause or the end of the study
Recurrence rate of hemoptysis | Every two months after treatment when the patient was assessed complete response; every month after treatment when assessed partial response, stable disease or progressive disease; up to progressive disease after the second treatment or within 36 months
  For the NSCLC subjects with hemoptysis, the patients completely or almost completely hemostasis were treated with the first treatment of DEB-BACE. If hemoptysis occurs during follow-up, it is recurrent of hemoptysis
Tumor biomarker (CEA, SCC) | Every two months after treatment when the patient was assessed complete response; every month after treatment when assessed partial response, stable disease or progressive disease; up to progressive disease after the second treatment or within 36 months
  Changes of tumor biomarkers
Quality of life score (EORTC, QLQ-30) | Every two months after treatment when the patient was assessed complete response; every month after treatment when assessed partial response, stable disease or progressive disease; up to progressive disease after the second treatment or within 36 months
  Changes of quality of life score; using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-30) Scores
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score (ECOG PS) | Every two months after treatment when the patient was assessed complete response; every month after treatment when assessed partial response, stable disease or progressive disease; up to progressive disease after the second treatment or within 36 months
  Changes of ECOG PS
VAS pain grade | Every two months after treatment when the patient was assessed complete response; every month after treatment when assessed partial response, stable disease or progressive disease; up to progressive disease after the second treatment or within 36 months
  Changes of VAS pain grade